CLINICAL TRIAL: NCT02291666
Title: Effects of Type 2 Diabetes on CYP450s Activities; Intersubject Variability in Drug Metabolism.
Brief Title: Evaluation of CYP450 Activities in Diabetic Patients vs. Non-diabetic Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CE 14.066
Record Dates: First submitted 2014-10-30; First posted 2014-11-14 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes
Keywords: Cytochromes p450; drug metabolism; pharmacokinetics; diabetes; probe markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Omeprazole; Caffeine; Wuc protein, Drosophila; Bupropion; Dextromethorphan; Midazolam; Tolbutamide; Chlorzoxazone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T2D patients with A1C ≤7.0 (Experimental): CRCHUM-MT cocktail; a single oral dose of the CRCHUM-MT cocktail will be administered; 100mg caffeine, 75mg bupropion, 150mg tolbutamide, 20mg omeprazole, 30mg dextromethorphan, 2mg midazolam and at night, one oral 250mg dose of chlorzoxazone will be taken separately.
  Interventions: Drug: CRCHUM-MT cocktail
- T2D patients with A1C>7.0 (Experimental): CRCHUM-MT cocktail; a single oral dose of the CRCHUM-MT cocktail will be administered; 100mg caffeine, 75mg bupropion, 150mg tolbutamide, 20mg omeprazole, 30mg dextromethorphan, 2mg midazolam and at night, one oral 250mg dose of chlorzoxazone will be taken separately.
  Interventions: Drug: CRCHUM-MT cocktail
- Non T2D subjects (Active Comparator): CRCHUM-MT cocktail; a single oral dose of the CRCHUM-MT cocktail will be administered; 100mg caffeine, 75mg bupropion, 150mg tolbutamide, 20mg omeprazole, 30mg dextromethorphan, 2mg midazolam and at night, one oral 250mg dose of chlorzoxazone will be taken separately.
  Interventions: Drug: CRCHUM-MT cocktail

INTERVENTIONS:
Drug: CRCHUM-MT cocktail
  Other Names: omeprazole; Losec; caffeine; Wake-up; bupropion; Wellbutrin; Zyban; dextromethorphan; midazolam; tolbutamide; chlorzoxazone; Acetazone

SUMMARY:
Type 2 diabetes (T2D) could modulate CYP450 activities involved in drug-metabolism and cardiovascular homeostasis. We propose to carry out, for the first time, a comprehensive characterization of the effects of T2D on the expression and activity of major CYP450s. In our studies, patients with T2D will be studied since hyperglycaemia and/or hyperinsulinemia are believed to modulate CYP450s. This vicious cycle puts patients at risk of micro- and macro-vascular complications and inadequately controlled T2D due to high intersubject variability in drug disposition and action.

Characterization of the effects of T2D on drug metabolism capacity will be performed using a cocktail of CYP450 probe drugs.

CYP450 phenotype will be determined in 3 groups of patients (n=126 patients): 1) 42 T2D patients with good glycemic control; 2) 42 T2D patients with poor glycemic control; and 3) 42 non-T2D healthy subjects following a single oral administration of a cocktail of CYP450 probe drugs. Subjects will receive the CRCHUM-MT cocktail consisting of caffeine (CYP1A2), bupropion (CYP2B6), tolbutamide (CYP2C9), omeprazole (CYP2C19), dextromethorphan (CYP2D6), midazolam (CYP3A4/5) and chlorxozaxone (which will be administered separately) (CYP2E1). Serial blood samples will be drawn and urine collected. Metabolic ratios will be calculated and compared between three groups of subjects. Other co-variables to be studied include T2D biomarkers at baseline (glucose, insulin, HbA1c), medications, genetic polymorphisms and inflammatory markers.

Our cocktail probe drug approach should allow us to demonstrate the effects of T2D on the activity of major CYP450s. Moreover, this project will indicate to us whether glycemic control should be considered as a covariate of intersubject variability in drug metabolism capacity.

DETAILED DESCRIPTION:
Patients with type 2 diabetes (T2D) require various therapeutic approaches (diet, exercise and drugs) to ensure glycaemic control while minimizing the risk of hypoglycaemia. T2D is also associated with vascular morbidities necessitating multiple drugs to prevent cardiovascular complications. Clinical practice reveals that T2D patients show highly variable responses to different drugs. Variable drug dosages and effects are observed for drugs such as clopidogrel, warfarin, cyclosporine and tacrolimus, as well as for anti-hypertensive, cholesterol lowering and antidiabetic drugs. These observations strongly suggest that T2D modulates factors regulating drug disposition and/or drug effects.

The hypothesis underlying this proposal is: T2D and its abnormalities alter the expression and activities of CYP450s involved in the disposition of drugs used to treat T2D and associated comorbidities.

The overall objective of this project is to investigate the effects of T2D on the activity of several CYP450 isozymes. Primary objective: To compare CYP450 activities between diabetic and non-diabetic subjects following a single oral administration of a cocktail of CYP450 probe drugs. The secondary objective: To evaluate and compare CYP450 activities according to the glycemic control (T2D patients with good glycemic control; T2D patients with poor glycemic control; and non-diabetic healthy subjects).

Study design; Patients (n=126) will be recruited to constitute 3 groups: Group I, 42 confirmed T2D with HbA1c ≤7.0; Group II, 42 patients with poor glycemic control HbA1c>7.0, and Group III, 42 sexed-matched non-T2D healthy subjects. This design will allow us to compare CYP450 activities between T2D patients with good glycemic control, T2D patients with poor glycemic control, and non-diabetic healthy subjects. Participants will be ≥18 years old, with a body weight index ≤35, and be non-smokers (>3 months). Subjects will be recruited at the CHUM outpatient clinic. The T2D diagnosis will be established according to the Canadian clinical guidelines. After an overnight fast, participants will be admitted to the CRCHUM's Clinical Research Unit (they will be not hospitalized). Subjects will receive the CRCHUM-MT cocktail; 100mg caffeine, 100mg bupropion, 250mg tolbutamide, 20mg omeprazole, 30mg dextromethorphan and 2mg midazolam to phenotype for CYP1A2, 2B6, 2C9, 2C19, 2B6, 2D6 and 3A4/5, respectively. Serial blood samples will be drawn and urine collected over 8 hours following drug administration. At the end of study day, subjects will be discharged from the CRCHUM's Clinical Research Unit and an oral 250mg dose of chlorzoxazone (CYP2E1) will be given and urine collected overnight for 12 hours.

A blood sample will be taken for pharmacogenetic analysis for relevant drug metabolizing enzymes. Additional blood samples will be collected just before the administration of the cocktail to measure insulin, glycaemia and HbA1c levels, biomarkers and inflammatory markers.

The subjects will be instructed not to take any medication, caffeine or theobromine containing products on the morning of study day. Their regular medication will be administered 4 hours after the administration of the cocktail if indicated. The subjects in whom our probe marker drugs are used daily will still be enrolled as metabolic ratios and will be determined to establish CYP450 activities.

Pharmacokinetic parameters such as oral clearance, metabolic clearance and renal clearance will be determined by noncompartmental analysis. Metabolic ratios will be calculated and compared between three groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥18 years old
* Body weight index ≤35,
* Non-smokers (>3 months)
* Patients with type 2 diabetes and good glycemic control (A1C<7) or poor glycemic control (A1C>7.0) and healthy non-diabetic subjects will be eligible.

Exclusion Criteria:

* Subjects with estimated glomerular filtration (MDRD) <50mL/min/1.73m2
* ALT and AST 3 times above the upper limit of normal
* Organ transplant recipient, inflammatory illnesses (i.e., polyarthritis, severe cirrhosis, infectious diseases, heart failure, HIV, hepatitis)
* Previous history of or an active cancer (except non-melanoma skin cancer)
* Uncontrolled thyroid functions
* Pregnant
* History of drug or alcohol abuse
* Subjects with a history of or current inflammatory bowel diseases including ulcerous colitis and Crohn's disease, and bariatric surgery
* Drugs known to modulate CYP450 activities, subject taking one of the following therapies will be excluded: antibiotics, antivirals, anticancers, CYP450 inducers (carbamazepine, phenobarbital, phenytoin, rifampin, St-John's wort), CYP450 inhibitors (amiodarone, fluvoxamine, fluoxetine, verapamil), immunosuppressors, warfarin, INFs, antibodies or grapefruit juice (<2-4 weeks) , CYP450 drugs with strong affinity for the selected isoform and with a long half-life, CYP450 mechanism-based inhibitors or an investigational drug
* Intolerance or hypersensitivity to probe drugs in the CRCHUM-MT cocktail or chlorzoxazone/acetaminophen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Metabolic ratio | 12 hours
  The metabolite/probe-drug (parent compound) ratio will be used as a metabolic index of CYP activity.

SECONDARY OUTCOMES:
Oral clearance | 12 hours
  CLo will be determined by noncompartmental analysis
Renal clearance | 12 hours
  CLr will be determined by noncompartmental analysis (Ae0-t of compound/AUC0-t compound)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, BPharm, PhD, Principal Investigator — Centre de recherche du Centre Hospitalier de l'université de Montréal (CHUM); Jean-Louis Chiasson, MD, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Gravel S, Chiasson JL, Turgeon J, Grangeon A, Michaud V. Modulation of CYP450 Activities in Patients With Type 2 Diabetes. Clin Pharmacol Ther. 2019 Dec;106(6):1280-1289. doi: 10.1002/cpt.1496. Epub 2019 Jul 9. PMID 31099895
- [Derived] Gravel S, Chiasson JL, Dallaire S, Turgeon J, Michaud V. Evaluating the impact of type 2 diabetes mellitus on CYP450 metabolic activities: protocol for a case-control pharmacokinetic study. BMJ Open. 2018 Feb 8;8(2):e020922. doi: 10.1136/bmjopen-2017-020922. PMID 29439084